CLINICAL TRIAL: NCT07327905
Title: Intravenous Lidocaine Infusion Versus Intravenous Dexmedetomidine Infusion During Laparoscopic Sleeve Gastrectomy : the Effect on Recovery Outcomes Variables
Brief Title: Intravenous Lidocaine Infusion Versus Intravenous Dexmedetomidine Infusion During Sleeve Gastrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, sarah mohamed, lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 0109246
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Bariatric Surgery; Lidocaine; Dexmedetomidine
Keywords: lidocaine; dexmedetomidine; bariatric

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group L (Active Comparator): receive lidocaine infusion
  Interventions: Other: intravenous lidocaine
- group D (Active Comparator): receive dexmedetomidine infusion
  Interventions: Other: intravenous dexmedetomidine

INTERVENTIONS:
Other: intravenous lidocaine — 20 patients will receive lidocaine infusion
  Other Names: group L
  Arms: group L
Other: intravenous dexmedetomidine — 20 patients will receive dexmedetomidine infusion
  Other Names: group D
  Arms: group D

SUMMARY:
Although laparoscopic (LAP) bariatric surgery is minimally invasive. Following any laparoscopic procedure, patients typically experience the peak of postoperative pain within the first 24 hours. This intense pain gradually subsides, with significant relief usually occurring by the 2nd or 3rd postoperative day. The initial peak and subsequent decline in pain intensity highlight the importance of effective early pain management strategies to ensure patient comfort and recovery during this critical period. Inadequate management of postoperative pain can result in serious complications. Lidocaine is increasingly recognised as a vital adjunct in managing perioperative pain. Its efficacy extends beyond traditional local anaesthetic applications, as it also demonstrates analgesic, anti-hyperalgesic, and anti-inflammatory properties. Dexmedetomidine is a highly selective alpha-2 adrenergic agonist with hypnotic, sedative, anxiolytic, sympatholytic, and analgesic effects, while causing minimal respiratory depression

DETAILED DESCRIPTION:
Morbid obesity is often linked to conditions such as diabetes, coronary artery disease, hypertension, hyperlipidaemia, and certain types of cancer, all of which negatively affect patients' quality of life, increase mortality risk, and shorten life expectancy. (1) Evidence suggests that medical approaches for weight loss, such as dietary therapy, physical activity, and behavioural modifications, typically do not lead to significant or sustained weight loss. In contrast, bariatric surgery is far more effective when combined with regular exercise and lifestyle changes. It remains the most successful and durable treatment for severe obesity and its related conditions, reducing the risk of 5-year mortality and significantly improving quality of life. (2) Laparoscopic sleeve gastrectomy has become a popular bariatric procedure due to its relative simplicity compared to more complex surgeries, such as gastric bypass or the full biliopancreatic diversion with duodenal switch (BPD/DS). The procedure can be performed laparoscopically, which is minimally invasive, leading to shorter recovery times and fewer complications. (3-5) Although laparoscopic (LAP) bariatric surgery is minimally invasive. Following any laparoscopic procedure, patients typically experience the peak of postoperative pain within the first 24 hours. This intense pain gradually subsides, with significant relief usually occurring by the 2nd or 3rd postoperative day. The initial peak and subsequent decline in pain intensity highlight the importance of effective early pain management strategies to ensure patient comfort and recovery during this critical period. Inadequate management of postoperative pain can result in serious complications, including delayed wound healing, impaired gastrointestinal function, myocardial ischaemia, immunologic changes, pulmonary issues, and an increased risk of thromboembolism due to immobility. (6) Centrally acting opioids have long been the cornerstone for managing severe postoperative pain. However, growing awareness of their side effects has sparked increasing interest in opioid-sparing multimodal analgesic strategies. This approach is particularly important in morbidly obese patients, who often present with multiple co-morbidities and face specific challenges related to anaesthesia and surgery. Opioid-sparing strategies in these patients not only aim to manage pain effectively but also minimise the risks associated with opioid use, improving overall postoperative outcomes. (7) Lidocaine is increasingly recognised as a vital adjunct in managing perioperative pain. Its efficacy extends beyond traditional local anaesthetic applications, as it also demonstrates analgesic, anti-hyperalgesic, and anti-inflammatory properties. By employing intravenous lidocaine infusions during the perioperative period, healthcare providers can enhance pain control, particularly in populations such as bariatric patients. Lidocaine achieves its effects through various mechanisms, including sodium channel blockade and inhibition of G protein-coupled receptors and N-methyl-D-aspartate (NMDA) receptors. This multifaceted action makes lidocaine a valuable component in multimodal analgesic regimens, ultimately improving patient comfort and recovery outcomes. (8,9) Dexmedetomidine is a highly selective alpha-2 adrenergic agonist with hypnotic, sedative, anxiolytic, sympatholytic, and analgesic effects, while causing minimal respiratory depression. Its sympatholytic properties lower mean arterial blood pressure (MAP) and heart rate (HR) by inhibiting the release of norepinephrine. Additionally, dexmedetomidine can reduce the need for both anaesthetic and opioid analgesics during the perioperative period. (10-13) AIM OF THE WORK The present study aims to evaluate the effect of intraoperative intravenous infusion of lidocaine versus intravenous infusion of dexmedetomidine on postoperative analgesia and opioid requirements.

The primary outcomes:

• Quality of pain control assessed by the visual analogue scale (VAS) in the first 24 hours after surgery at rest and at movement.

The secondary outcomes:

* The total amount of rescue opioids administered in the first 24 hours post-operatively. (mg).
* Time until the first analgesic requirement. (hours).
* Duration of stay in the PACU. (hours).
* Patients' satisfaction score.
* The incidence of post-operative complications, such as nausea, vomiting, and hypoxaemia.

PATIENTS

Study settings:

The present study will be conducted in the Alexandria Main University Hospital.

Study design:

The study will be prospective, randomised, double-blinded: The anaesthesiologist, the patient, and the outcome assessor will be unaware of the group allocation. An independent anaesthesiologist will prepare the study drugs.

Sample size calculation:

The sample size is determined according to the recommendation of the Department of Statistics, Medical Research Institute, Alexandria University.

Power Analysis Table N1 N2 Actual Powerb Test Assumptions Power Std. Dev1 Std. Dev2 Mean Difference Sig. Test for Mean Differencea 20 20 .806 .8 .9 .7 .740 .05

1. Two-sided test.
2. Based on noncentral t-distribution. By using SPSS program version 28, (14) A minimal total sample size of (40) patients with laparoscopic sleeve gastrectomy (20) per group is needed to detect an assumed difference of (0.74) (15,16) in mean visual analogue scale (VAS) between a group of patients receiving intraoperative intravenous infusion of lidocaine vs another group receiving intravenous infusion of dexmedetomidine with assumed group SDs of (0.9,0.7) respectively to evaluate the effect of both procedures regarding quality of pain control in the first 2 hours after surgery using independent t test with a significance level of (0.05) and 80% power.

Study population:

All patients will be randomly assigned 1:1 using a sealed envelope method. Patients will be categorised randomly into two equal groups; both groups will undergo laparoscopic sleeve gastrectomy under general anaesthesia and receive paragastric autonomic neural blockade with the administration of:

Group L: Intravenous lidocaine. Group D: Intravenous dexmedetomidine.

METHODS

Preoperative evaluation and preparation:

* During the preoperative visit, evaluation of patients will be carried out through proper history taking, clinical examination and routine laboratory investigations including complete blood picture, coagulation profile, blood urea, serum creatinine and any other necessary investigations.
* Informed written consent will be obtained from all patients included in the study during the preoperative visit.
* Patients will be trained on a visual analogue scale, with 0 corresponding to no pain and 10 to the worst pain imaginable.
* Patients will be informed about the analgesic regimen.
* Thrombotic prophylaxis (enoxaparin 40 mg) will be started 12 hours before surgery.

The assigned study drugs preparation

The independent anaesthesiologist not involved in any other aspect of the included patient's care will prepare the different blinded solutions and code them:

Loading Dose:

* Group L: Loading dose of lidocaine at 1.5 mg kg-1 (with a maximum dose of 100 mg).
* Group D: Loading dose of dexmedetomidine at 0.5 µg kg-1. Both will be diluted in 250 cc of normal saline.

Maintenance dose:

* Group L: 400 mg of lidocaine will be diluted in a 50 cc syringe infusion pump containing normal saline, achieving a concentration of 8 mg ml-1.
* Group D: 100 μg of dexmedetomidine will be diluted in a 50 cc syringe infusion pump containing normal saline, achieving a concentration of 2 μg ml-1.

Monitoring

On arrival to the operative theatre, an intravenous cannula will be inserted and standard monitoring will be established using a multichannel monitor (Carescape Monitor B650, GE Healthcare Finland) to monitor the following in both groups:

* Electrocardiogram (ECG) for heart rate and rhythm (Beats/min).
* Non-invasive measurement of arterial blood pressure (Mean blood pressure in mmHg).
* Peripheral oxygen saturation (SpO2%).
* End tidal CO2 tension (in mmHg).
* Nerve Stimulator.
* Temperature probe. Anaesthetic management Participants will be categorised randomly into two groups: Group L and Group D. Patients in both groups will receive the loading dose of their assigned study drugs during the 10 minutes preceding the induction of anaesthesia. Following this, the syringes containing the maintenance dose will be infused at a rate of 0.25 ml kg-1 hr-1 for both groups, corresponding to doses of 2 mg kg-1 hr-1 for lidocaine and 0.5 µg kg-1 hr-1 for dexmedetomidine.

After preoxygenation for 3 minutes, anaesthesia will be induced in both groups with propofol 2 mg kg-1 until loss of verbal response, fentanyl 2 µg kg-1. Endotracheal intubation will be facilitated by intravenously injecting rocuronium 0.6 mg kg-1. Anaesthesia will be maintained by isoflurane with 50% oxygen in air (1.2-1.5 %) to maintain entropy between 40-60, and a capnogram will be attached. Mechanical ventilation settings will include volume-controlled mode with a tidal volume of 6 - 8 ml kg-1 and a respiratory rate of 12-15 cycles min-1 to maintain an end-tidal carbon dioxide tension between 35 and 40 mmHg and an oxygen saturation of ≥ 95%. Incremental doses of rocuronium will be guided by nerve stimulator (TOF), 0.15-0.25 indicates adequate surgical relaxation.

All drug doses calculated in mg kg-1 were based on the patients' ideal body weight. (17)

All patients will receive:

* Paracetamol 1 g.
* Dexamethasone 8 mg.
* Diclofenac 75 mg.
* Ondansetron 4 mg.
* Magnesium 2.5 g. Patients in both groups will receive a paragastric autonomic neural blockade after establishing pneumoperitoneum.

Technique of paragastric autonomic neural blockade:

The paragastric lesser omentum neural block will be performed by the surgeon using a 25-gauge short needle connected to a venous catheter extension, introduced through the left 12-mm port. The needle will be capped during insertion and will be uncapped inside the abdomen using a grasper, ensuring it remains under direct visualisation at all times. A total of 20 ml of plain 0.5% bupivacaine will be injected at six levels within the fatty tissue of the paragastric region, with careful aspiration before each injection to prevent inadvertent blood vessel injection. The anaesthetic will be carefully administered along the lesser omentum, targeting the vagus nerve and its distal branches at the esophagogastric junction, proximal stomach, mid-stomach, and distal antrum. The hepatic artery area will then be infiltrated, followed by the left gastric artery in the posterosuperior paragastric region by lifting the proximal half of the sleeve from the stomach's neo-greater curvature. After the infiltration is complete, the needle will be recapped and removed from the abdominal cavity.

The infusion of intravenous lidocaine and intravenous dexmedetomidine syringes will be stopped upon completion of the surgical methylene blue test.

Recruitment manoeuvres will be conducted at least twice during surgery: once after induction and again before the patient is awakened.

All intravenous and inhaled medications will be discontinued after skin closure is completed. At the end of the operation, the oxygen flow will be adjusted to 6 L min-1. Neuromuscular blockade will be reversed with sugammadex 2 mg kg1. All patients will be extubated when they meet the criteria for extubation in the operating room before their transfer to the post-anaesthesia care unit (PACU).

Postoperative care:

Postoperatively, all patients will be assessed for the presence and severity of pain using the Visual Analogue Scale at PACU arrival and in the ward for the first 24 hours and will be recorded at 30 minutes, 2, 6, 12, 18, and 24 hours.

In both groups, postoperative analgesia consisted of:

* Paracetamol (1 g per 6 h).
* Diclofenac (75 mg every 12 h for the first 2 postoperative days). In addition, a rescue dose of IV Nalbuphine 4 mg per bolus will be administered if VAS is ≥ 4 and will be repeated every 30 minutes until VAS is less than 4.

Patients will be discharged from the PACU when an Aldrete score > 9 (18) is achieved. Health care providers in the PACU and ward will be blinded to patient group assignment and to the nature of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-50 years, both sexes.
* American Standards Association (ASA) physical status class II to III.
* Body mass index (BMI) 35-50 kg m-².

Exclusion Criteria:

* Cardiac conduction disorders.
* Cardiomyopathy.
* Chronic opioid use.
* Allergy to the studied medications.
* Pregnancy and breastfeeding.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-26 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale | postoperative day 1
  at rest , movement

SECONDARY OUTCOMES:
time to first nalbuphine dose | postoperative day 1
  minutes
patient satisfaction | postoperative day1
  • Poor = 1, fair = 2, good = 3, excellent = 4.
postoperative nalbuphine requirements | postoperative day 1
  mg
postoperative complications | postoperative day 1
  nausea , vomiting

CONTACTS AND LOCATIONS:
Overall Officials: sarah m elgamal, MD, Principal Investigator — Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh V, Pahade A, Mowar A. Comparing Efficacy of Intravenous Dexmedetomidine and Lidocaine on Perioperative Analgesic Consumption in Patients Undergoing Laparoscopic Surgery. Anesth Essays Res. 2022 Jul-Sep;16(3):353-359. doi: 10.4103/aer.aer_121_22. Epub 2022 Dec 9. PMID 36620103